CLINICAL TRIAL: NCT05541575
Title: Discussion on Virtual Reality Intervention Course: Exploring the Effectiveness of the Attitude of Care
Brief Title: Exploring the Effectiveness the Attitude, Competence of Care, Empathy Among the Home Care Workers With Dementia People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, PhD, RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FJU-C109203
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Empathy; Attitude; Competence
Keywords: home caregivers, careers
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Experimental: offered 3 films of VR course of BPSD for 30 mins to each participants.
  Interventions: Other: VR films
- No intervention (No Intervention): NO films of VR course of BPSD to any participants.

INTERVENTIONS:
Other: VR films — A new virtual reality course for home care workers to experience the view of dementia people with BPSD and the relative feelings.
  Arms: Intervention

SUMMARY:
This study develop a new virtual reality course for home care workers to experience the view of dementia people with BPSD and the relative feelings. After the intervention, the experimental group would completed the several scales of attitude of care, competence of care and empathy, then the factor analysis and correlation analysis were measured.

In the first stage, a single group pre and post test study was conducted to extract 10 home caregivers of dementia care from Hondao Senior Citizen's Welfare Foundation. In order to explore the VR course affect the attitude of care, competent of care and empathy towards the dementia people in community, and future career.

In the second stage, this study use quasi experimental design. The experimental group (n=65) and the control group (n=65) each have a pre- and post-test design. The experimental group uses virtual reality courses for intervention experience, while the control group does not have intervention. After the two post-tests are completed, then provide the same immersive 3D VR experience as the experimental group. The measurement tools in this study used the Jefferson Empathy Scale (Chinese Version), The Interpersonal Reactivity Index (Chinese Version), and three self-made scales focus on dementia care attitude scale, the dementia care competency scale and the virtual reality course experience scale.

DETAILED DESCRIPTION:
More than 90% of people with mild and moderate level of dementia live at home in the community. The behaviors and psychological symptoms of dementia (BPSD) would be severe by age, and often increases the difficulty and pressure for family caregivers. Also the outcome from the relative studies are limited.

This study develop a new virtual reality course for home care workers to experience the view of dementia people with BPSD and the relative feelings. After the intervention, the experimental group would completed the several scales of attitude of care, competence of care and empathy, then the factor analysis and correlation analysis were measured.

In the first stage, a single group pre and post test study was conducted to extract 10 home caregivers of dementia care from Hondao Senior Citizen's Welfare Foundation. In order to explore the VR course affect the attitude of care, competent of care and empathy towards the dementia people in community, and future career.

In the second stage, this study use quasi experimental design. The experimental group (n=65) and the control group (n=65) each have a pre- and post-test design. The experimental group uses virtual reality courses for intervention experience, while the control group does not have intervention. After the two post-tests are completed, then provide the same immersive 3D VR experience as the experimental group. The measurement tools in this study used three self-made scales focus on dementia care attitude scale, the dementia care competency scale and the virtual reality course experience scale and empathy scale. ANCOVA would be used for the correlation analysis above scales.

Home care workers can use VR as an appropriate interventions, to empathize with the situation, faced and recognize the weakness, frustration and emotional distress of dementia people. Then change the attitude and arise the competency of care, also should be considered for ensure that patients with dementia stay in good care quality.

ELIGIBILITY:
Inclusion Criteria:

1. is currently or has been serving as an in-home caregiver for a community-dwelling patient with dementia;
2. aged 20 years and above
3. conversant in Mandarin and Taiwanese
4. agreed to participate in this study

Exclusion Criteria:

1. age 19 years and below
2. disagreed to participate in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Empathy Scale | Change from Baseline, T1
  It contains 9 questions. There is no subscale. The score of range from 1-5.
Dementia care scale | Change from Baseline, T1
  It contains 22 questions. There is 3 subscale. The score of range from 1-5.
Virtual reality course experience scale | Experimental group need to completion 30 mins intervention, then participants fill the questionnaire.
  It contains 9 questions. There is 3 subscale. The score of range from 1-5.

SECONDARY OUTCOMES:
Empathy Scale | Through study completion, an average of 2 months(T2)
  It contains 9 questions. There is no subscale. The score of range from 1-5.
Dementia care scale | Through study completion, an average of 2 months(T2)
  It contains 22 questions. There is 3 subscale. The score of range from 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Hsieh, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Fooyin University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollock M, Hornabrook RW. The prevalence, natural history and dementia of Parkinson's disease. Brain. 1966 Sep;89(3):429-48. doi: 10.1093/brain/89.3.429. No abstract available. PMID 5921126
- [Background] Elliott R, Bohart AC, Watson JC, Greenberg LS. Empathy. Psychotherapy (Chic). 2011 Mar;48(1):43-9. doi: 10.1037/a0022187. PMID 21401273
- [Background] Hattink B, Meiland F, van der Roest H, Kevern P, Abiuso F, Bengtsson J, Giuliano A, Duca A, Sanders J, Basnett F, Nugent C, Kingston P, Droes RM. Web-Based STAR E-Learning Course Increases Empathy and Understanding in Dementia Caregivers: Results from a Randomized Controlled Trial in the Netherlands and the United Kingdom. J Med Internet Res. 2015 Oct 30;17(10):e241. doi: 10.2196/jmir.4025. PMID 26519106
- [Background] Wijma EM, Veerbeek MA, Prins M, Pot AM, Willemse BM. A virtual reality intervention to improve the understanding and empathy for people with dementia in informal caregivers: results of a pilot study. Aging Ment Health. 2018 Sep;22(9):1115-1123. doi: 10.1080/13607863.2017.1348470. Epub 2017 Jul 10. PMID 28691861
- [Background] Dyer E, Swartzlander BJ, Gugliucci MR. Using virtual reality in medical education to teach empathy. J Med Libr Assoc. 2018 Oct;106(4):498-500. doi: 10.5195/jmla.2018.518. Epub 2018 Oct 1. PMID 30271295
- [Background] Shin D. Empathy and embodied experience in virtual environment: To what extent can virtual reality stimulate empathy and embodied experience? Comput Hum Behav. 2018;78:64-73. doi:10.1016/j.chb.2017.09.012
- [Background] Jutten LH, Mark RE, Maria Janssen BWJ, Rietsema J, Droes RM, Sitskoorn MM. Testing the effectivity of the mixed virtual reality training Into D'mentia for informal caregivers of people with dementia: protocol for a longitudinal, quasi-experimental study. BMJ Open. 2017 Aug 21;7(8):e015702. doi: 10.1136/bmjopen-2016-015702. PMID 28827242
- [Background] Jutten LH, Mark RE, Sitskoorn MM. Can the Mixed Virtual Reality Simulator Into D'mentia Enhance Empathy and Understanding and Decrease Burden in Informal Dementia Caregivers? Dement Geriatr Cogn Dis Extra. 2018 Dec 6;8(3):453-466. doi: 10.1159/000494660. eCollection 2018 Sep-Dec. PMID 30631337
- [Background] Sari DW, Igarashi A, Takaoka M, Yamahana R, Noguchi-Watanabe M, Teramoto C, Yamamoto-Mitani N. Virtual reality program to develop dementia-friendly communities in Japan. Australas J Ageing. 2020 Sep;39(3):e352-e359. doi: 10.1111/ajag.12797. Epub 2020 Jun 2. PMID 32483931
- [Background] Kim D. Development and Effect of Virtual Reality Practice Program for Improving Practical Competency of Caregivers Specializing in Dementia. Healthcare (Basel). 2021 Oct 18;9(10):1390. doi: 10.3390/healthcare9101390. PMID 34683070